CLINICAL TRIAL: NCT06433531
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Efficacy of TQH2929 in Healthy Adult Subjects and Psoriasis Subjects
Brief Title: A Clinical Study of TQH2929 Injection in Treatment With Generalized Pustular Psoriasis (GPP)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQH2929-I-01 (Ib)
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQH2929 Injection (900 mg) (Experimental): TQH2929 Injection is administered as a single dose.
  Interventions: Drug: TQH2929 Injection

INTERVENTIONS:
Drug: TQH2929 Injection — TQH2929 injection is a humanized monoclonal antibody that interfering with the signal cascade.

SUMMARY:
This study is a multicenter, single-group, open-label study to evaluate the safety and tolerability of TQH2929 injection at a dose of 900mg in adult subjects with active Generalized Pustular Psoriasis (GPP), and to preliminarily evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 75 years (inclusive)，both male and female；
* A known and documented history of Generalized Pustular Psoriasis diagnosed with European Rare and Severe Psoriasis Expert Network (ERASPEN) criteria in 2017；
* Presenting with a moderate-severe flare of Generalized Pustular Psoriasis (GPP)
* Body mass index (BMI) within 18~36 kg/m2；
* Major organ function is good;
* Patients must be able to understand and sign a written informed consent document;
* Patients must be able to complete study-related procedures and questionnaires;
* Female and male subjects of childbearing age should agree to use contraceptive measures during the study period and within 6 months after the end of the study; Female subjects need to serum pregnancy pregnancy test within 7 days before study enrollment.

Exclusion Criteria:

* Patients with primary plaque psoriasis vulgaris with pustules that are restricted to psoriatic plaques；
* Immediate life-threatening flare of Generalized Pustular Psoriasis or requiring intensive care treatment, according, to the judgment of the investigator；
* Computed Tomography of the chest shows active or occult tuberculosis or a history of contact with an open tuberculosis (TB) subject within the past 6 months. Subjects positive for tuber closes spot(T-SPOT) (or other tuberculosis diagnostic test) result;
* Active hepatitis during the screening period, or positive for hepatitis B surface antigen (HBsAg)；
* History of human immunodeficiency virus (HIV) infection, or positive HIV serological results at screening during screening；
* Positive antibodies to treponema pallidum during screening；
* History of serious infection leading to hospitalization or intravenous infusion of antibiotics or antiviral therapy within 3 months prior to baseline;
* Active systemic infections requiring systemic antibiotics or systemic antiviral therapy within 4 weeks prior to baseline;
* History of opportunistic infection and parasitic infection within 6 months prior to the screening period；
* History of herpes zoster infection within 2 months prior to baseline；
* Subject has known or suspected autoimmune disease;
* Receive major surgery within 4 weeks prior to the first dose;
* Subjects with any type of active malignancy or a history of malignancy (except cervical cancer or non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma and papillary thyroid carcinoma) that has been cured for more than 5 years prior to the screening period;
* Subjects have history of significant drug allergies；
* Use of the following medications within the prescribed time:

  1. Receive topical drugs for the treatment of skin diseases within 1 weeks prior to baseline;
  2. Receive systemic therapy within 4 weeks prior to baseline;
  3. Receive regular phototherapy within 4 weeks prior to baseline;
  4. Within 12 weeks prior to baseline, receive live (attenuated) vaccine;
  5. Receive antibiotics and antivirals within 4 weeks prior to baseline.
* People who are alcoholic, drug addicts, and known drug dependents;
* Pregnant or Breasting feeding subject;
* Received a blood transfusion within 4 weeks prior to the first dose;
* Subject is unable to tolerate intravenous infusion administration;
* During the period of participation in this study, participants had planned surgical procedures;
* Have participated in clinical trials of other drugs or medical devices within 4 weeks prior to baseline;
* In the judgment of the investigator or sponsoring medical auditor, it is believed that there are any medical or psychiatric symptoms that put the subject at risk, interfere with participation in the study, or interfere with the interpretation of the results of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | From the first dose to 113 days after the last dose
  The occurrence of all adverse events (AE).
Serious adverse events (SAE) | From the first dose to 113 days after the last dose
  The occurrence of all serious adverse events (SAE).
Treatment-related adverse events(TRAE) | From the first dose to 113 days after the last dose
  The occurrence of all treatment-related adverse events(TRAE).
Clinical laboratory abnormalities | From the first dose to 113 days after the last dose
  Incidence of participants with clinical laboratory abnormalities

SECONDARY OUTCOMES:
Time to reach maximum observed serum concentration (Tmax) | Single dose: within 1 hour (pre-dose), 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours post-dose
  Time to reach maximum (peak) serum concentration following drug administration.
Maximum serum concentration (Cmax) | Single dose: within 1 hour (pre-dose), 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours post-dose
  The Cmax is the maximum observed serum concentration of study drug.
Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) | Single dose: within 1 hour (pre-dose), 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours post-dose
  Area under the concentration-time curve of the TQH2929 Injection in serum over the time interval from 0 extrapolated to infinity.
Area Under the Concentration-Time Curve From 0 to Last Observation (AUC [0-t]) | Single dose: within 1 hour (pre-dose), 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours post-dose
  Area under the concentration-time curve of the TQH2929 Injection in serum over the time interval from 0 extrapolated to the last quantifiable data point.
Apparent volume of distribution (Vd/F) | Single dose: within 1 hour (pre-dose), 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours post-dose
  Apparent volume of distribution of the TQH2929 Injection in serum.
Apparent clearance (CL/F) | Single dose: within 1 hour (pre-dose), 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours post-dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Half-life (t1/2) | Single dose: within 1 hour (pre-dose), 0, 0.5, 1, 2, 6, 12, 24, 48, 72, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2016, 2353, 2688 hours post-dose
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the serum.
Anti-drug antibodies (ADA) | Single dose: within 1 hour (pre-dose), Days 15, 57, 85, and 113 post-dose
  A participant was considered ADA-positive across the study if they had a positive reading at any time point during the study.
Proportion of patients with a generalized pustular psoriasis physician global assessment (GPPGA) pustulation subscore of 0/1 at Weeks 1,2,4 | 1, 2 and 4 weeks post-dose
  The Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) relies on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The investigator (or qualified site personnel) scored the erythema, pustules, and scaling of all GPP lesions from 0 to 4. A lower GPPGA pustulation subscore indicates a better outcome. A GPPGA pustulation subscore of 0 means no visible pustules. The proportion of patients who achieved a GPPGA pustulation subscore of 0/1 at Week 1,2,4 is reported.
Percent change in generalized pustular psoriasis area and severity index (GPPASI) from baseline at weeks 1,2,4 | Baseline and 1,2,4 weeks post-dose
  GPPASI provides a numeric scoring for a patient's overall Generalized Pustular Psoriasis (GPP) disease state, ranging from 0 (no disease) to 72 (worse disease state). It is a linear combination of percent of surface area of skin affected by erythema, pustules, and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions (head, trunk, upper limbs and lower limbs).
Proportion of patients with a generalized pustular psoriasis physician global assessment (GPPGA) score of 0 or 1 at week 1 | Baseline and 1,2,4 weeks post-dose
  GPPGA relied on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The GPPGA total score was calculated by taking the mean of the erythema subscore, pustules subscore and scaling/crusting subscore. The severity of each subscore was assessed using a 5 point scale score ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe).
  A lower GPPGA score indicates a better outcome, with 0 being clear and 1 being almost clear. The proportion of patients with a GPPGA score of 0 or 1 at Week 1,2,4 is reported.
Change in generalized pustular psoriasis area and severity index (GPPASI) from baseline at week 1,2,4. | Baseline and 1,2,4 weeks post-dose
  Generalized Pustular Psoriasis Area and Severity Index (GPPASI) provides a numeric scoring for a patient's overall Generalized Pustular Psoriasis (GPP) disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin affected by erythema, pustules, and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions (head, trunk, upper limbs and lower limbs). A higher score indicates a worse disease state, while a score of 0 indicates no disease.
Change from baseline in psoriasis symptom scale (PSS) score at week 1,2,4 | Baseline and 1,2,4 weeks post-dose
  PSS is a 4-item patient-reported outcome instrument that assesses the severity of psoriasis symptoms in moderate to severe psoriasis patients. The symptoms included are: pain, redness, itching, and burning. The symptom severity was assessed using a 5 point scale ranging from 0 to 4 where 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe. The symptom scores are added to an unweighted total score (range: 0 to 16). A lower PSS score indicates a better outcome.
Proportion of patients with psoriasis symptom scale (PSS) score of 0 at week 1,2,4. | 1,2,4 weeks post-dose
  PSS is a 4-item patient-reported outcome instrument that assesses the severity of psoriasis symptoms in moderate to severe psoriasis patients. The symptoms included are: pain, redness, itching, and burning. The symptom severity was assessed using a 5 point scale ranging from 0 to 4 where 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe.
Change from baseline in dermatology life quality index (DLQI) score at weeks 1,2,4 | Baseline and 1,2,4 weeks post-dose.
  The DLQI is a 10-item questionnaire that asks participants to evaluate the degree that their skin problem has affected their quality of life in the last week in the following 6 aspects: symptoms and feelings, daily activities, leisure, work or school activities, personal relationships and treatment related feelings. Participants answer the 10 questions on a scale from 0 (not at all) to 3 (very much). The DLQI is calculated by summing the scores of the 10 questions, resulting in a maximum of 30 and a minimum of 0 with higher scores indicating more impaired quality of life. A negative change from Baseline indicates improvement.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical Universitye, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Second People's Hospital of Chengdu, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang